CLINICAL TRIAL: NCT00660868
Title: Agapurin Retard Used in Patients With Smell Disorder- A Post-marketing Observational Study
Brief Title: Is Pentoxifylline Able to Improve Olfactory Sensitivity?
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK157072007
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Olfaction Disorders
Keywords: smell; olfaction; olfactory sensitivity; smell loss; chemoreception
MeSH Terms: conditions — Olfaction Disorders; Anosmia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with posttraumatic, idiopathic, and postinflammatory cause of smell loss; patients age between 18 and 50 years. Odor threshold better than 1.
  Interventions: Drug: Pentoxifylline retard 400mg

INTERVENTIONS:
Drug: Pentoxifylline retard 400mg — Agapurin retard 400mg 3/day per os for 3 weeks
  Other Names: Agapurin retard

SUMMARY:
Signal processing in the olfactory neuron could be influenced by inhibition of enzymes like phosphodiesterase. Pentoxifylline is a unspecific phosphodiesterase inhibitor. The hypothesis is that pentoxifylline could lead to increased sensitivity to odors.

DETAILED DESCRIPTION:
Olfactory signal processing is conducted by a G-protein linked increase of intracellular concentration of adenosine 3´,5´-cyclic monophosphate (cAMP). In the cilia of olfactory sensory neurons (OSN) cAMP is degraded by phosphodiesterase 1C2 (PDE1C2). Inhibition of PDE1C2 could result in an increased response of OSN to chemical stimuli. Aim of the present prospective post-marketing surveillance study was to investigate the impact of pentoxifylline, an unspecific phosphodieasterase inhibitor, on olfactory function.

ELIGIBILITY:
Inclusion Criteria:

* hyposmic or functionally anosmic patients TDI-score <31
* age: 18-50 years
* odor threshold: better than 1
* cause of smell loss: post traumatic, postinflammatory, idiopathic

Exclusion Criteria:

* normosmic patients,
* patients with contraindications for application of pentoxifylline
* patients that cannot give written agreement to the study
* patients under 18 years and over 50 years of age

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: hyposmic or functionally anosmic patients TDI-score <31; age: 18-50 years; odor threshold: better than 1; cause of smell loss: post traumatic, postinflammatory, idiopathic
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
TDI-score | at day 0 and follow up after 3 weeks

SECONDARY OUTCOMES:
odor threshold odor discrimination odor identification | at day 0 and at follow up after 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Volker Gudziol, Dr. med., Principal Investigator — Technische Universität Dresden
Locations (1):
- Zentrum für Riechen und Schmecken, Universitäts- HNO- Klinik Dresden, Dresden, Germany